CLINICAL TRIAL: NCT06936176
Title: A Prospective, Multicenter, Single-Arm Objective Performance Criteria Clinical Trial Evaluating the Safety and Efficacy of a Single-Use Neurovascular Intravascular Shockwave Catheter and Intravascular Shockwave Therapy Device for Pretreatment of Calcified Lesions in the Extracranial Carotid Artery (CREATE Trial)）
Brief Title: Prospective Trial of IVL for Calcified Carotid Lesions(CREATE Trial)
Acronym: CREATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Bluesail Boyuan Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LFBY-202501
Record Dates: First submitted 2025-04-12; First posted 2025-04-20 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Carotid Artery Stenosis
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with calcified extracranial carotid artery stenosis (Experimental): Study Arm: Single-arm, prospective, multicenter trial evaluating the safety and efficacy of the Neurovascular Intravascular Shockwave Catheter and Intravascular Shockwave Therapy Device for pretreatment of calcified lesions in the extracranial carotid artery prior to carotid artery stenting (CAS).
  Interventions: Device: Neurovascular Intravascular Shockwave Catheter

INTERVENTIONS:
Device: Neurovascular Intravascular Shockwave Catheter — Device:
  Neurovascular Intravascular Shockwave Catheter (single-use, rapid-exchange balloon catheter with integrated shockwave emitters).
  Intravascular Shockwave Therapy Device (IVL-HVG-N01, generates localized shockwaves to fracture calcifications).
  Procedure:
  Patients undergo standard CAS preparation with guidewire placement and cerebral protection.
  If conventional balloon angioplasty fails (residual stenosis >70%), the IVL catheter is advanced to the target lesion.
  Shockwave therapy is applied at 6 atm, followed by low-pressure balloon dilation (8 atm) if needed.
  Subsequent stent deployment is performed per standard practice.

SUMMARY:
* Clinical Trial Summary

  * Trial Title:** CREATE Trial: Safety and Efficacy of IVL for Carotid Calcified Lesions
  * Sponsor:** Shanghai Bluesail Boyuan Medical Technology Co., Ltd.
  * Clinical Trial Leader:** Beijing Anzhen Hospital
  * Coordinating Investigator:** Prof. Huo Xiaochuan
* Study Purpose This trial assesses a new device-a single-use neurovascular intravascular shockwave catheter and therapy device-for treating calcified blockages in the carotid artery. It uses sound waves to break up calcium deposits, facilitating stent placement and blood flow restoration.
* Eligibility

  * Adults aged 18-80 with severe carotid artery narrowing (≥50% symptomatic or ≥70% asymptomatic) due to calcium buildup.
  * Patients who failed standard balloon dilation.
  * Exclusions include pregnancy, recent strokes/heart attacks, uncontrolled hypertension, or other high-risk conditions.
* Study Design

  * **Type:** Prospective, multicenter, single-arm trial.
  * **Sample Size:** 204 patients across multiple hospitals.
  * **Duration:** 1-month follow-up post-procedure.
* Procedures

  1. **Pre-treatment:** Imaging (CT angiography, ultrasound) to confirm eligibility.
  2. **Procedure:** Shockwave catheter breaks up calcium, followed by stent placement.
  3. **Follow-up:** Assessments at 7 days (or discharge) and 1 month post-procedure.
* Benefits and Risks

  * **Benefits:** Improved stent placement success, reduced risk of complications, minimally invasive with shorter recovery time.
  * **Risks:** Bleeding, infection, vessel damage, stroke, heart attack, device malfunction. Risks are closely monitored with emergency protocols.
* Patient Protections

  * Ethics committee approval and strict safety guidelines.
  * Voluntary participation with the option to withdraw anytime.
  * Free treatment and compensation for trial-related injuries.
* For Healthcare Providers

  * **Innovation:** Adapts coronary lithotripsy technology for carotid use.
  * **Evidence:** Supported by preclinical data and a pilot study (100% success rate in 5 patients).
  * **Endpoints:** Primary: Stent success (residual stenosis <30%) and 30-day major adverse events. Secondary: Device success rate, repeat procedures, long-term outcomes.
* Contact Information

For questions, contact:

**Ms. Zhang Yanjiao** Email: yanjiao.zhang@jwmsgrp.com

DETAILED DESCRIPTION:
**Detailed Clinical Trial Description**

### **1. Background and Rationale** **Clinical Need:**

* **Carotid artery calcification** is a major contributor to ischemic stroke, accounting for 15-20% of cases. Severe calcification complicates stent placement, leading to high rates of residual stenosis and adverse events (e.g., stroke, myocardial infarction) with conventional treatments like balloon angioplasty.
* **Current Limitations:** Standard therapies often fail to adequately modify calcified plaques, necessitating high-pressure balloon dilation, which risks embolization, vessel dissection, or hemodynamic instability.

**Innovative Solution:**

* The **intravascular lithotripsy (IVL) system** delivers localized sonic pressure waves to fracture calcium deposits while sparing soft tissue, enabling safer stent deployment.
* **Evidence Base:** Supported by coronary IVL trials (e.g., DISRUPT CAD I-IV) and off-label carotid case reports demonstrating 90-100% technical success with minimal complications.

  ### **2. Study Objectives** **Primary Objectives:**
* **Efficacy:** Assess **surgical success rate** (stent placement with residual stenosis <30%).
* **Safety:** Evaluate **30-day major adverse events (MAE)** (composite of death, stroke, or myocardial infarction).

**Secondary Objectives:**

* Device success rate (successful delivery/retrieval of IVL catheter).
* Rates of target lesion revascularization, ipsilateral stroke, and MACCE (major adverse cardiac/cerebrovascular events).

  ### **3. Methodology** **Study Design:**
* **Prospective, multicenter, single-arm, objective performance criteria (OPC) trial.**
* **No control group** due to ethical concerns (standard therapy failure is an inclusion criterion).

**Intervention:**

1. **IVL Catheter:** Rapid-exchange balloon catheter with integrated electrodes generating sonic waves (80 pulses max per device).
2. **IVL Device:** Console delivering controlled energy pulses (compatible with 3.0-5.0 mm balloons).

**Procedure Steps:**

* **Pre-treatment:** Dual antiplatelet therapy (aspirin + clopidogrel) for ≥3 days.
* **IVL Delivery:**
* Balloon inflation to 6 atm, followed by 10 pulses/cycle (up to 8 cycles).
* Stent placement post-calcium modification.
* **Post-procedure:** Monitoring for MAE at 7 days and 1 month.

**Key Assessments:**

* **Imaging:** CT angiography (baseline), DSA (intraoperative), ultrasound (follow-up).
* **Clinical:** NIHSS/mRS scores, vital signs, lab tests (hematology, biochemistry).

  * **4. Participant Selection** **Inclusion Criteria:**
* Symptomatic (≥50%) or asymptomatic (≥70%) carotid stenosis with circumferential calcium >50% (CTA-confirmed).
* Failed conventional balloon pre-dilation (residual stenosis >70%).
* Modified Rankin Scale (mRS) score ≤2.

**Exclusion Criteria:**

* Vulnerable plaques, recent stroke/MI (within 2-12 weeks), or contraindications to antiplatelets.
* Severe comorbidities (e.g., NYHA Class IV heart failure, creatinine >2.5 mg/dL).

  ### **5. Risk Management** **Anticipated Risks:**
* **Procedure-related:** Vessel dissection (1-3%), embolic stroke (2-5%), access-site hematoma.
* **Device-related:** Balloon rupture, electrode malfunction (<1%).

**Mitigation Strategies:**

* **Embolic protection devices** mandatory.
* **Strict operator training** (≥5 supervised cases required).
* **Real-time monitoring** for hemodynamic instability (bradycardia/hypotension).

  ### **6. Statistical Plan** **Sample Size Justification:**
* **Efficacy endpoint:** 107 patients needed (95% expected vs. 85% OPC, α=0.025, power=90%).
* **Safety endpoint:** 204 patients (4.5% expected vs. 11% OPC).
* **Total:** 204 (accounting for 10% dropout).

**Analysis Populations:**

* **Full Analysis Set (FAS):** All treated patients (intent-to-treat).
* **Per-Protocol Set (PPS):** Excludes major protocol deviations.

**Statistical Tests:**

* Primary endpoints: **One-sided 95% CI** (success rate lower bound >85%; MAE upper bound <11%).
* Secondary endpoints: Descriptive statistics (rates, Kaplan-Meier survival analysis).

  ### **7. Ethical and Regulatory Compliance**
* **Ethics Approval:** Obtained from all site IRBs (reference: LFBY-202501).
* **Informed Consent:** Mandatory, with provisions for legally authorized representatives.
* **Data Protection:** Compliant with China's Personal Information Protection Law (PIPL).

  ### **8. Operational Oversight**
* **Monitoring:** Centralized EDC (Medidata Rave) with 100% source data verification.
* **Audits:** Independent DSMB reviews safety data biannually.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years (inclusive), gender unrestricted.
2. Extracranial carotid artery: Preoperative CT angiography (CTA) confirms symptomatic carotid stenosis ≥50% or asymptomatic carotid stenosis ≥70% with calcification (CTA measurement: calcification > 50% of circumference).

   Note: (Extracranial carotid artery: Internal carotid artery or carotid bifurcation; Symptomatic refers to having had a non-disabling ischemic stroke or TIA within 6 months.)
3. Intraoperative digital subtraction angiography (DSA) confirms carotid stenosis ≥50% (by NASCET criteria) or asymptomatic carotid stenosis ≥70% (by NASCET criteria).
4. Participants with a pre-enrollment modified Rankin Scale (mRS) score ≤2.
5. Participants planned for carotid artery stenting (CAS) who have failed conventional balloon dilation.
6. Patients or their legal guardians understand the purpose of the trial, provide informed consent, and agree to follow-up.

Exclusion Criteria:

1. Target lesion caused by non-atherosclerotic disease.
2. Participants with complete occlusion of the target lesion or contralateral carotid artery.
3. Participants with severe disability due to cerebral infarction.
4. Participants with large acute or subacute thrombi near the target lesion, or with arteriovenous malformations or aneurysms.
5. Participants with tortuous target lesion vessels that prevent stent placement.
6. Participants with symptomatic severe stenosis in other cerebral vessels.
7. Participants requiring concurrent or additional surgical interventions during the trial period.
8. Participants with tandem severe stenosis or occlusion in vessels proximal or distal to the target lesion.
9. Participants who have had a myocardial infarction or large cerebral infarction within 2 weeks prior to screening.
10. Participants who have had intracranial hemorrhage within 3 months prior to screening.
11. Participants with vulnerable or high-risk plaques (unstable, prone to rupture, and thrombosis leading to acute cardiovascular events or death) as judged by carotid ultrasound.
12. Participants with uncontrolled hypertension (systolic blood pressure persistently ≥180 mmHg or diastolic blood pressure persistently ≥110 mmHg).
13. Participants with known platelet count < 90×10^9/L, severe liver impairment (transaminases > 3 times the upper limit of normal), severe renal impairment (serum creatinine > 2.5 mg/dL [221 µmol/L]), or New York Heart Association Class IV heart failure.
14. Participants with coagulopathy (INR ≥2.0) or contraindications to heparin or antiplatelet agents.
15. Participants with active infections.
16. Participants unable to use cerebral protection devices.
17. Participants allergic to components of the investigational device or contrast agents (excluding rash).
18. Participants with life expectancy less than 1 year.
19. Pregnant or breastfeeding women.
20. Participants currently enrolled in another drug or medical device clinical trial (before reaching the primary endpoint).
21. Other situations where the investigator deems the participant unsuitable for the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Procedural Success Rate | Immediately post-procedure (intraoperative).
  Successful stent deployment with residual stenosis <30% after the procedure (via angiography).
30-Day Major Adverse Events (MAE) Rate | 30 days (±7 days) post-procedure.
  Composite of:
  All-cause death； Stroke (ischemic or hemorrhagic, with neurological deficits lasting ≥24h)； Myocardial infarction (MI) (per standard diagnostic criteria).

SECONDARY OUTCOMES:
Device Success | Intraoperative
  Successful delivery, activation, and retrieval of the neurovascular intravascular shockwave (IVL) catheter without technical failure.
Device Malfunction Rate | Intraoperative
  The Device Malfunction Rate is the percentage of procedures where the IVL catheter or device fails to operate as intended, including issues like balloon rupture or electrode malfunction.
Target Lesion Revascularization Rate | Within 7 days/Before Discharge, 1 Month Postoperative
  The incidence of revascularization treatment for the initially treated lesion vessel after surgery.
Ipsilateral Stroke Rate | Within 7 days/Before Discharge, 1 Month Postoperative
  The occurrence of a stroke event on the same side as the target vessel in the subject.
Major Adverse Cardio-Cerebrovascular Events (MACCE) Rate | Within 7 days/Before Discharge, 1 Month Postoperative
  A composite of all-cause death, any stroke, any myocardial infarction, and any revascularization.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing An Zhen Hospital of the Capital University of Medical Sciences, Beijing, China